CLINICAL TRIAL: NCT06804798
Title: Evaluation of Catheter Associated Urinary Tract Infection Between Metal Alloy Coated Catheter and Conventional Latex Catheter in Critically Ill Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National University of Malaysia (Other)
Responsible Party: Principal Investigator, Mohammad Nizam Mokhtar, Dr, National University of Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FF-2023-056
Record Dates: First submitted 2025-01-17; First posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Sepsis; Urosepsis; Intensive Care Unit
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Intervention Model Description: The interventional study is between urinary catheter and conventional latex urinary catheter and metal alloy coated urinary catheter
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional latex urinary catheter (Active Comparator)
  Interventions: Device: Latex metal alloy coated catheter
- Latex metal alloy coated catheter (Experimental)
  Interventions: Device: conventional latex urinary catheter

INTERVENTIONS:
Device: Latex metal alloy coated catheter — Metal alloy works as an antiseptic whereby preventing the attachment of biofilm to the catheter lining.
  Arms: Conventional latex urinary catheter
Device: conventional latex urinary catheter — Latex catheters prove to be soft, flexible, inexpensive and thermo-sensitive towards body temperature. However, there is a risk of developing CAUTI as bacteria are more susceptible to adhere to latex.
  Arms: Latex metal alloy coated catheter

SUMMARY:
This is a prospective single blinded randomized trial to evaluate the incidence of catheter associated urinary tract infection (CAUTI) between latex catheter and metal alloy coated catheter among Intensive Care Unit (ICU) patients. CAUTI has a few definitions, in this study, we will follow the latest Central of Disease Control (CDC) guideline definition of CAUTI in January 2022.

This study involves 100 patients who meet the inclusion and exclusion criteria that have been set. The patients will be divided into group A and group B and two types of catheters will be given out to the healthcare workers according to the randomization. Data collection involves demographic, medical and laboratory data and will be documented in the tables provided. All data will be collected from day of urinary catheterization in ICU until patients discharge or die or maximum of 14 days in ICU or develop CAUTI or ABUTI or whichever that occurred earlier. Patients who died within 48 hours of catheter insertion, will be considered as drop-out.

Data that has been extrapolated from this study will then give us an insight regarding the best type of catheter to avoid CAUTI, risk factors associated with CAUTI and to determine length of ICU stay and ICU morbidity with patients who have CAUTI. This study proves to be important in reducing the overall healthcare associated infection in the ICU setting.

ELIGIBILITY:
Inclusion criteria

1. Adult more than 18 years old
2. Indwelling urinary catheter more than 48 hours Exclusion Criteria

1. Community urosepsis 2. Chronic kidney disease and end stage renal failure 3. Suprapubic catheter 4. Patient with dependent urinary catheter 5. Pregnant ladies 6. Congenital urinary tract abnormality 7. Surgical procedure involving urinary tract 8. Moribound patient or expected to die within 24 hours 9. Discharged to ward within 48 hours 10. Latex allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
To Compare | 2 years
  To compare catheter associated urinary tract infections rate between conventional latex urinary catheter and latex metal alloy

SECONDARY OUTCOMES:
To compare | 2 years
  To compare the rate of bacteremia from catheter associated urinary tract infection between conventional latex urinary catheter and latex metal alloy catheter
To compare | 2 years
  To compare the common types of microorganisms associated with catheter associated urinary tract infection between conventional latex urinary catheter and latex metal alloy catheter
To compare | 2 years
  To compare risk factor that is associated with catheter associated urinary tract infection between conventional latex urinary catheter and latex metal alloy catheter
To compare | 2 years
  To compare the incidence of acute kidney injury (AKI) in catheter associated urinary tract infection between conventional latex urinary catheter and latex metal alloy catheter
Length of stay | 2 years
  To determine length of stay in ICU and ICU mortality in catheter associated urinary tract infection between conventional latex urinary catheter and latex metal alloy catheter

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Canselor Tuanku Muhriz, Universiti Kebangsaan Malaysia, Bandar Tun Razak, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided